CLINICAL TRIAL: NCT01185327
Title: Do Isreali Infants of Ethiopian Origin Mother Regurgitate More Than Other Infants?
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Erez Nadir, MD, Hillel Yaffe medical center
Other Study IDs: 0066-10-HYMC-CTIL
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Rumination
Keywords: Regurgitation; Infants to Israeli Ethiopian-origin mothers
MeSH Terms: conditions — Rumination Syndrome; Gastroesophageal Reflux | interventions — Lactation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study: Infants to Israeli Ethiopian-origin Mothers
  Interventions: Behavioral: Breastfeeding
- Control: Infants to Israeli non-Ethiopian-origin mothers
  Interventions: Behavioral: Breastfeeding

INTERVENTIONS:
Behavioral: Breastfeeding — Breastfeeding

SUMMARY:
Nursing team of well baby nursery at Hillel Yaffe medical center in Hadera, Israel have noticed that infant of Ethiopian-origin mothers regurgitate more than other infants. Probably, these infants are breastfeed much more than other infants.

Some Ethiopian-origin mothers are used to eat teff-flower porridge during the last weeks of pregnancy and after birth, in order to expand milk production.

Study goal is to find out if infants of Ethiopian-origin mother do regurgitate more than others, and if they weight gain is similar to other infants. Another goal is to find out if breastfeeding mothers of Ethiopian origin do eat that porridge, and if there is any difference between those who do eat that porridge and those who do not.

DETAILED DESCRIPTION:
Nursing team of well baby nursery at Hillel Yaffe medical center in Hadera, Israel have noticed that infant of Ethiopian-origin mothers regurgitate more than other infants. Probably, these infants are breastfeed much more than other infants.

Some Ethiopian-origin mothers are used to eat teff-flower porridge during the last weeks of pregnancy and after birth, in order to expand milk production.

Study goal is to find out if infants of Ethiopian-origin mother do regurgitate more than others, and if they weight gain is similar to other infants. Another goal is to find out if breastfeeding mothers of Ethiopian origin do eat that porridge, and if there is any difference between those who do eat that porridge and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at Hillel Yaffe medical center during 2009 (To Ethiopian origin mother in study group, and to non-Ethiopian origin mothers in control group)

Exclusion Criteria:

* Infants who were transferred to NICU for any reason.

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants born at Hillel Yaffe medical center during 2009
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
% weight decrease | First week of life
  Proportion of minimal weight during hospitalization to birth weight

SECONDARY OUTCOMES:
Number of regurgitations per day | First week of life

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe medical center, Hadera, Israel
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

REFERENCES:
- [Background] Barak M, Lahav S, Mimouni FB, Dollberg S. The prevalence of regurgitations in the first 2 days of life in human milk- and formula-fed term infants. Breastfeed Med. 2006 Autumn;1(3):168-71. doi: 10.1089/bfm.2006.1.168. PMID 17661594
- [Background] Hegar B, Dewanti NR, Kadim M, Alatas S, Firmansyah A, Vandenplas Y. Natural evolution of regurgitation in healthy infants. Acta Paediatr. 2009 Jul;98(7):1189-93. doi: 10.1111/j.1651-2227.2009.01306.x. Epub 2009 Apr 21. PMID 19397533
- [Background] Asefa M, Hewison J, Drewett R. Traditional nutritional and surgical practices and their effects on the growth of infants in south-west Ethiopia. Paediatr Perinat Epidemiol. 1998 Apr;12(2):182-98. doi: 10.1046/j.1365-3016.1998.00104.x. PMID 9620568
- [Background] Wenlock RJ, Wenlock RW. Maternal nutrition, prolonged lactation and birth spacing in Ethiopia. J Biosoc Sci. 1981 Jul;13(3):261-8. doi: 10.1017/s0021932000013456. PMID 7276029
- [Background] Getahun Z, Scherbaum V, Taffese Y, Teshome B, Biesalski HK. Breastfeeding in Tigray and Gonder, Ethiopia, with special reference to exclusive/almost exclusive breastfeeding beyond six months. Breastfeed Rev. 2004 Nov;12(3):8-16. PMID 17891858
- [Background] Meftuh AB, Tapsoba LP, Lamounier JA. Breastfeeding practices in Ethiopian women in southern California. Indian J Pediatr. 1991 May-Jun;58(3):349-56. doi: 10.1007/BF02754966. PMID 1937647
- [Background] Zeisel SH. Is maternal diet supplementation beneficial? Optimal development of infant depends on mother's diet. Am J Clin Nutr. 2009 Feb;89(2):685S-7S. doi: 10.3945/ajcn.2008.26811F. Epub 2008 Dec 30. PMID 19116319